CLINICAL TRIAL: NCT00966108
Title: Evaluation of SENSIMED Triggerfish for 24 Hour IOP Monitoring in Healthy Subjects and Glaucoma Patients
Brief Title: SENSIMED Triggerfish Discomfort During IOP Monitoring
Acronym: 09/02
Status: Completed | Type: Observational
Sponsor: Sensimed AG (Industry)
Responsible Party: Prof. Dr. med. Norbert Pfeiffer, Universitätsmedizin der Johannes Gutenberg-Universität Mainz
Other Study IDs: 09/02
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Safety and Tolerability of SENSIMED Triggerfish in Glaucoma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy subjects
  Interventions: Device: SENSIMED Triggerfish
- Glaucoma patients
  Interventions: Device: SENSIMED Triggerfish

INTERVENTIONS:
Device: SENSIMED Triggerfish — Ocular Telemetry Sensor for IOP monitoring

SUMMARY:
Evaluation of the wearing discomfort (safety and tolerability) involved during IOP monitoring with the SENISMED Triggerfish, a sensor embedded in a telemetric contact lens

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to comply with the study procedure
* Patient is 18-80 years old
* Healthy subject or glaucoma patient
* Patient has consented to be in the trial and signed informed consent is available before any study related procedures are carried out
* Cylinder refraction of no more than +/- 2 diopters in the study eye
* Visual acuity of 20/80 or better in the study eye
* Ability of subject to understand the character and individual consequences of the study
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Subjects wearing contact lenses within the last two years
* Subjects with contraindications for wearing contact lenses
* History of refractive surgery
* History of intraocular surgery in the last three months
* Severe dry eye syndrome
* Keratoconus or other corneal abnormalities
* Conjunctival or intraocular inflammation
* Pregnancy and lactation
* Simultaneous participation in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects and glaucoma patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
ocular discomfort on a visual analogue scale | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Pfeiffer, Prof. Dr. med., Principal Investigator — Universitätsmedizin Mainz
Locations (1):
- Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate, Germany